CLINICAL TRIAL: NCT06153394
Title: Prolonged Hypercoagulability Following Major Liver Resection for Malignancy
Acronym: PRIORITY
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: Valeo Pharma Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 123658
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Hepatic Disease; Surgery-Complications; Hypercoagulability; Thrombosis
MeSH Terms: conditions — Digestive System Diseases; Thrombophilia; Thrombosis | interventions — enoxaparin sodium; Injections; Dalteparin

STUDY DESIGN:
Intervention Model Description: This will be a phase III pilot trial where 50 participants will be randomized 1:1 to receive extended duration thromboprophylaxis via Redesca or standard of care thromboprophylaxis via Fragmin. Participants will be followed for 3 years after surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Redesca (Experimental): Patients in the extended thromboprophylaxis group will receive Redesca (enoxaparin sodium for injection) (40mg) once a day, starting on the day of surgery, for 90 days postoperatively.
  Interventions: Drug: Redesca (enoxaparin sodium for injection)
- Fragmin (Active Comparator): Patients in the standard of care group will receive Fragmin (daletparin) (5,000 I.U) once a day, starting on the day or surgery, for 30 days postoperatively.
  Interventions: Drug: Fragmin (dalteparin)

INTERVENTIONS:
Drug: Redesca (enoxaparin sodium for injection) — Redesca is low molecular weight heparin and a biosimilar biologic drug (biosimilar) to Lovenox. Indications have been granted on the basis of similarity between Redesca and the reference biologic drug Lovenox. As such, Redesca (enoxaparin sodium) is indicated for thromboprophylaxis in patients undergoing high risk abdominal and colorectal surgeries. Doses are provided as self-administered subcutaneous injections using a pre-filled syringe with a protective shield.
  Arms: Redesca
Drug: Fragmin (dalteparin) — Fragmin is a low molecular weight heparin indicated for thromboprophylaxis in patients undergoing high risk abdominal and colorectal surgeries. Doses are provided as self-administered subcutaneous injections using a pre-filled syringe with a protective shield. Our institution uses this drug for standard of care thromboprophylaxis (30 days) in this patient population.
  Arms: Fragmin

SUMMARY:
This clinical trial will investigate the ability of thromboelastrogrpahy (TEG®) to detect hypercoagulability after liver surgery and will examine the effect of extended thromboprophylaxis (medical treatment to prevent the development of blood clots inside blood vessels) in patients undergoing liver surgery for cancer treatment.

The liver plays a key role in regulating the process of blood clotting. As a result, blood clots are a major cause of complications and death following liver surgery. This is especially true in cancer patients who are at a higher risk of developing blood clots. Current methods for preventing clotting complications after liver surgery include conventional coagulation blood tests (CCTs) and anticoagulant drugs, such as low molecular weight heparins (LMWHs). Current LMWH treatment is prescribed for one month after surgery, but studies show that the risk of developing blood clots can last up to 3 months. Studies also show that CCTs may not be as effective in detecting clotting issues as more comprehensive testing systems, such as TEG. This study will randomize 50 participants to receive 90 days of thromboprophylaxis (using the LMWH Redesca) or the standard of care 30 days (using the LMWH Fragmin) after liver surgery. The medication will be given by injection, similar to a regular vaccine or an insulin injection. Participants will inject the medication every day, for 30 or 90 days, after surgery. Participants will also have their blood tested for clotting issues via TEG testing before surgery and on post-operative days 1,3,5,30 and 90. After surgery, participants will be monitored by their surgeon for clotting complications and 3 year disease-free survival.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older at the time of enrollment.
2. Requiring major liver resection (>2 liver sections) for any oncologic indication.
3. Requiring postoperative thromboprophylaxis will be included.
4. Willing and able to perform subcutaneous injections according to the study protocol, or receive injections form a caregiver delegated by the participant.

Exclusion Criteria:

1. Anyone below 18 years of age.
2. Patients on current anticoagulant and/or antiplatelet therapy
3. Patients with a history of thrombotic events
4. Patients with a coagulation disorder.
5. Patients with recognized thrombophilia.
6. Patients who cannot understand/speak or read in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Number pf participants with hypercoagulability identified via TEG testing | Preoperatively (with pre-admission blood work) through to 90 days postoperatively
  All participants will have postoperative TEG testing performed for the detection of hypercoagulability.

SECONDARY OUTCOMES:
Thrombotic Events | Up to 6 months postoperatively
  Determining the occurrence of postoperative venous thrombotic events between treatment groups
Disease Free Survival | Up to 3 years postoperatively
  Comparing disease free survival (DFS) rates between treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Anton Skaro, MD PhD, Principal Investigator — Western Univeristy/LHSC
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Not planning to share IPD with other researchers